CLINICAL TRIAL: NCT04495218
Title: Implementation of a Next-generation Sequencing Analysis of a Panel of Genes Implicated in Incomplete Forms of Albinism
Brief Title: NGS Panel of Incomplete Forms of Ocular Albinism
Acronym: DIA
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2019/52
Record Dates: First submitted 2020-07-20; First posted 2020-07-31 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Albinism, Ocular
Keywords: Next generation sequencing; Albinism
MeSH Terms: conditions — Albinism, Ocular; Albinism | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patient with a diagnosis of incomplete form of albinism
  Interventions: Biological: Blood samples

INTERVENTIONS:
Biological: Blood samples — Performed a 10 ml blood sample (2 unnamed samples of 5ml) in each of the 100 patients included.

SUMMARY:
Implementation of a next-generation sequencing panel of genes to identify deleterious variants in patients with incomplete forms of albinism.

DETAILED DESCRIPTION:
Scientific context : Albinism is clinically characterised by cutaneous hypopigmentation and ophthalmologic features. These features common to all forms of albinism are foveal hypoplasia, misrouting of the optic nerves at the chiasm, retinal hypopigmentation, translucent irides and nystagmus. The molecular genetic lab at Bordeaux University Hospital is the national reference for the study of this disease. More than 1400 patients have been analyzed with a strategy including next-generation sequencing of the 19 known genes of albinism and array-CGH. Despite this thorough analysis, 25% of patients remain without molecular diagnosis. Our experience tells us that these patients often show an incomplete form of albinism with the presence of only few ophthalmologic signs. The molecular diagnosis is very challenging as the phenotype often overlaps with other ophthalmologic disorders.

ELIGIBILITY:
Inclusion Criteria:

* Minor and adult patient.
* Patient presenting a clinical diagnosis of incomplete form of albinism with presence of at least 2 signs of ocular albinism among which nystagmus, low vision, foveal hypoplasia, retinal hypopigmentation, translucent irides, misrouting of the optic nerves at the chiasm.
* Registered for the social security system.
* Informed consent signed by patient or parent of a minor patient.

Exclusion Criteria:

* Refusal to participate in research protocol.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with a clinical diagnosis of incomplete form of albinism with presence of at least 2 signs of ocular albinism among which nystagmus, low vision, foveal hypoplasia, retinal hypopigmentation, translucent irides, misrouting of the optic nerves at the chiasm and having a specialized consultation in CHU de Bordeaux
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Percentage of patients for whom a molecular diagnosis is obtained based on the panel of targeted genes | Enrollment
  the prevalence of finding at least two pathogenic variants is 10%.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Bordeaux, Bordeaux, France